CLINICAL TRIAL: NCT02644538
Title: A Randomized, Controlled, Open-label, Multicenter Clinical Trial to Evaluate the Addition of PegIFN Alfa-2a to CHB Patients Treated With Nucleot(s)Ides
Brief Title: Addition of PegIFN Alfa-2a to CHB Patients Treated With Nucleot(s)Ides
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Collaborators: People's Hospital of Anshun City of Guizhou Province (Other); The First Affiliated Hospital of Nanchang University (Other); First Affiliated Hospital of Xinjiang Medical University (Other)
Responsible Party: Principal Investigator, Peng Hu, Director of Department of infection disease, The Second Affiliated Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APACE
Record Dates: First submitted 2015-12-28; First posted 2016-01-01 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Hepatitis B
Keywords: HBsAg clearance
MeSH Terms: conditions — Hepatitis B | interventions — peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- nucleot(s)ides treated (No Intervention): patients who treated with nucleot(s)ides (including lamivudine, adefovir, entecavir, tenofovir) are still using the original treatment for 72 weeks
- PegIFN alfa-2a + nucleot(s)ides treated (Active Comparator): patients who treated with nucleot(s)ides (including lamivudine, adefovir, entecavir, tenofovir), then will add PegIFN alfa-2a to the original nucleot(s)ides for 48 weeks, then follow up for 24 weeks
  Interventions: Drug: PegIFN alfa-2a

INTERVENTIONS:
Drug: PegIFN alfa-2a — chronic hepatitis B patients who treated with nucleot(s)ides (including lamivudine, adefovir, entecavir, tenofovir) arrived HBV DNA <1000copies/ml, and HBsAg<3000IU/ml, then change the treatment to original nucleot(s)ides add on PegIFN alfa-2a, the combined treatment is for 48 weeks, and follow up for 24 weeks
  Other Names: Pegasys
  Arms: PegIFN alfa-2a + nucleot(s)ides treated

SUMMARY:
This study evaluates whether PegIFN alfa-2a add on can improve CHB patients HBsAg clearance at the end of 48 weeks treatment. The CHB patients who received nucleot(s)ides anti-virus treatment and reached HBV DNA<1000 copies/ml and HBsAg<3000 IU/ml, were randomly assigned into two groups: One group continue the nucleot(s)ides treatment for 72 weeks, the other add on PegIFN alfa-2a on the basis of the original treatment for 48 weeks, and follow up for 24 weeks.

DETAILED DESCRIPTION:
nucleot(s)ides is a potent inhibitor of hepatitis B viral(HBV) replication, but long-term therapy may be required, and it is difficult for CHB patients to achieve HBsAg clearance by using nucleot(s)ides. Therefore, it is need take long-term therapy if chronic hepatitis B (CHB) choose to use nucleot(s)ides, and in another way, nucleot(s)ides resistance is an important clinical risk. More and more young patients want to stop treating, and discontinuation of nucleot(s)ides is a feasible strategy to reduce resistance. However, it is really easy to relapse if patients did not arrive HBsAg clearance. PegIFN alfa-2a can clear HBV by direct anti-viral and immune regulation mechanisms including enhancing natural killer cell response, increased cluster of differentiation 8(CD8 +) T lymphocytes and other mechanisms to restore and enhance the immune response in patients with CHB; and what's more, patients are safety after discontinuing.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects,18-65 years
2. positive for hepatitis B surface antigen (HBsAg) and negative for antibodies to HBsAg (anti-HBs antibodies) for at least 6 months before NAs treated
3. nucleot(s)ides monotherapy (including lamivudine, adefovir, entecavir, tenofovir) and achieved HBV DNA<1000 copies/mL with HBsAg <3000 IU/mL, positive or negative for HBeAg, and negative for anti-HBs antibodies
4. Subjects with no contra-indications to Peginterferon alfa therapy as detailed in the label (Hypersensitivity to the active substance, to alpha interferon, or to any of the excipients; Autoimmune hepatitis; Severe hepatic dysfunction or decompensated cirrhosis of the liver; A history of severe pre-existing cardiac disease, including unstable or uncontrolled cardiac disease in the previous six months)
5. Subjects who are not co-infected with Hepatitis A Virus, Hepatitis C Virus or HIV
6. Female subjects not pregnant or breast feeding when Peginterferon alfa treatment commenced, and aware of the requirement to use an effective method of contraception during therapy
7. Written informed consent signed.

Exclusion Criteria:

1. positive for Hepatitis A Virus Ab, HCV-RNA or positive for Hepatitis C Virus Ab, HDV Ab, HEV Ab or positive for HIV Ab in screening period
2. Hepatocellular carcinoma(HCC) or alpha feto protein(AFP) levels more than 100 ng/ml and Hepatic malignant potential of Imaging examination or AFP levels more than 100 ng/ml for 3 months
3. Compensated or Decompensated liver cirrhosis: with history of cirrhosis before nucleot(s)ides treatment or Child-Pugh score ≥ 5 or Complications of liver cirrhosis such as ascites, hepatic encephalopathy, esophageal gastric varices bleeding
4. Autoimmune disease including Autoimmune hepatitis and Psoriasis and so on
5. Pregnant women and lactating women or patients with pregnancy plans and not willing to use contraception during the study period
6. A history of immunoregulation drug therapy within one year before entry including IFN and so on
7. Have a history of alcohol abuse
8. With severe psychiatric condition or nervous disease such as epilepsy, depression, mania, epilepsy, schizophrenia and so on
9. A neutrophil count of less than 1500 per cubic millimeter or a platelet count of less than 90,000 per cubic millimeter
10. Severe organ dysfunction
11. With other malignant tumors(exclude the cured ones)
12. Uncontrolled diabetes, hypertension or thyroid disease
13. A serum creatinine level that was more than 1.5 times the upper limit of the normal range
14. Hypersensitivity to interferon(IFN) or its active substance, and ineligible to IFN
15. Participate in other clinical studies at the same time
16. Patients unsuitable for the research -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants who achieve HBsAg clearance | treat for 48 weeks
  To investigate whether Peg-IFN alfa-2a add on treatment can improve the HBsAg clearance in CHB patients at the end of the treatment (48 week).

SECONDARY OUTCOMES:
Number of participants who achieve HBsAg seroconversion | 48 weeks
  To investigate whether Peg-IFN alfa-2a add on treatment can improve the HBsAg seroconversion in CHB patients at the end of the treatment (48 week).
Number of participants who achieve HBeAg clearance and seroconversion | 48 weeks
  To investigate whether Peg-IFN alfa-2a add on treatment can improve HBeAg clearance and seroconversion at the end of the treatment (48 week).
HBsAg changes from Baseline | 12,24 and 48 weeks
  Pegasys 24 weeks Group:12,24 weeks and Pegasys 48 weeks Group:12,24,48 weeks
Number of participants who achieve HBV DNA<1000 copies/ml | 12,24 and 48 weeks
  To investigate whether Peg-IFN alfa-2a add on treatment can improve HBV DNA<1000 copies/ml

IPD SHARING:
Plan to Share IPD: Undecided
still undecided

REFERENCES:
- [Result] Ganem D, Prince AM. Hepatitis B virus infection--natural history and clinical consequences. N Engl J Med. 2004 Mar 11;350(11):1118-29. doi: 10.1056/NEJMra031087. No abstract available. PMID 15014185
- [Result] Liang X, Bi S, Yang W, Wang L, Cui G, Cui F, Zhang Y, Liu J, Gong X, Chen Y, Wang F, Zheng H, Wang F, Guo J, Jia Z, Ma J, Wang H, Luo H, Li L, Jin S, Hadler SC, Wang Y. Epidemiological serosurvey of hepatitis B in China--declining HBV prevalence due to hepatitis B vaccination. Vaccine. 2009 Nov 5;27(47):6550-7. doi: 10.1016/j.vaccine.2009.08.048. Epub 2009 Sep 1. PMID 19729084
- [Result] Lu FM, Zhuang H. Management of hepatitis B in China. Chin Med J (Engl). 2009 Jan 5;122(1):3-4. No abstract available. PMID 19187608
- [Result] European Association For The Study Of The Liver. EASL clinical practice guidelines: Management of chronic hepatitis B virus infection. J Hepatol. 2012 Jul;57(1):167-85. doi: 10.1016/j.jhep.2012.02.010. Epub 2012 Mar 20. No abstract available. PMID 22436845
- [Result] Micco L, Peppa D, Loggi E, Schurich A, Jefferson L, Cursaro C, Panno AM, Bernardi M, Brander C, Bihl F, Andreone P, Maini MK. Differential boosting of innate and adaptive antiviral responses during pegylated-interferon-alpha therapy of chronic hepatitis B. J Hepatol. 2013 Feb;58(2):225-33. doi: 10.1016/j.jhep.2012.09.029. Epub 2012 Oct 6. PMID 23046671
- [Result] Chen J, Wang Y, Wu XJ, Li J, Hou FQ, Wang GQ. Pegylated interferon alpha-2b up-regulates specific CD8+ T cells in patients with chronic hepatitis B. World J Gastroenterol. 2010 Dec 28;16(48):6145-50. doi: 10.3748/wjg.v16.i48.6145. PMID 21182232
- [Result] Marcellin P, Bonino F, Yurdaydin C, Hadziyannis S, Moucari R, Kapprell HP, Rothe V, Popescu M, Brunetto MR. Hepatitis B surface antigen levels: association with 5-year response to peginterferon alfa-2a in hepatitis B e-antigen-negative patients. Hepatol Int. 2013 Mar;7(1):88-97. doi: 10.1007/s12072-012-9343-x. Epub 2012 Mar 23. PMID 23518903
- [Result] Piratvisuth T, Marcellin P, Popescu M, Kapprell HP, Rothe V, Lu ZM. Hepatitis B surface antigen: association with sustained response to peginterferon alfa-2a in hepatitis B e antigen-positive patients. Hepatol Int. 2013 Jun;7(2):429-36. doi: 10.1007/s12072-011-9280-0. Epub 2011 Jun 24. PMID 21701902
- [Result] Ning Q, Han M, Sun Y, Jiang J, Tan D, Hou J, Tang H, Sheng J, Zhao M. Switching from entecavir to PegIFN alfa-2a in patients with HBeAg-positive chronic hepatitis B: a randomised open-label trial (OSST trial). J Hepatol. 2014 Oct;61(4):777-84. doi: 10.1016/j.jhep.2014.05.044. Epub 2014 Jun 7. PMID 24915612